CLINICAL TRIAL: NCT02302248
Title: A Randomized, Active-Controlled Trial to Investigate the Effectiveness of a Crowdsourced Cognitive Reappraisal Intervention.
Brief Title: Effectiveness of a Crowdsourced Cognitive Reappraisal Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Collaborators: Northwestern University (Other); Columbia University (Other); University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1311006002
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crowdsourced Reappraisal (Experimental): Participants received the web-based crowdsourcing reappraisal intervention.
  Interventions: Behavioral: Crowdsourcing reappraisal intervention
- Expressive Writing (Active Comparator): Participants received the web-based expressive writing intervention.
  Interventions: Behavioral: Expressive writing intervention

INTERVENTIONS:
Behavioral: Crowdsourcing reappraisal intervention — 3 week access to a web-based crowdsourcing reappraisal platform.
  Arms: Crowdsourced Reappraisal
Behavioral: Expressive writing intervention — 3 week access to a web-based expressive writing platform.
  Arms: Expressive Writing

SUMMARY:
This study evaluates a web-based, crowdsourcing platform to promote cognitive reappraisal. Half of participants will be granted access to the crowdsourced reappraisal platform. The other half will be provided a web-based expressive writing platform. The investigators hypothesize that the crowdsourcing reappraisal platform will be more effective than the expressive writing platform in promoting positive psychological outcomes.

DETAILED DESCRIPTION:
There are many ways to manage stress and mood, including exercise, diet, and relaxation practices. Cognitive-based techniques are also extremely powerful. Simply changing how you think about stressful situations can dramatically affect the way you feel. Individuals who routinely use strategies like cognitive reappraisal exhibit an enviable affective profile: studies suggest these individuals generally have less stress, lower incidence of depression, and better social functioning than those who rely on less adaptive emotion regulatory techniques. Techniques like cognitive reappraisal are also integral to many evidence-based psychotherapeutic traditions, such as cognitive-behavioral therapy and rational-emotive therapy.

Unfortunately, cognitive techniques can be hard to learn. Thinking flexibly about stressful thoughts and situations requires creativity and poise, faculties that often elude us when we need them the most. In this study, the investigators evaluate a web-based technology that uses crowdsourcing and peer-to-peer interactions to help people learn cognitive-based techniques and apply them throughout their daily lives.

The goal of the proposed study is to see whether the investigators' technology is more engaging and more effective at reducing depression symptoms than a web-based expressive writing platform. While the investigators are most interested in how this intervention affects depression symptoms, the investigators will also assess other psychological variables and the investigators will open the study to the general population.

Participation in this study will last three weeks. Participants will be randomly assigned to receive either a crowdsourcing reappraisal platform or an expressive writing platform. All study procedures (subject recruitment, baseline and follow-up assessments, interventions) will be conducted online.

ELIGIBILITY:
Inclusion Criteria:

* An email account, a desktop computer, and broadband Internet access
* Access to modern web browsers (e.g., Chrome, Safari, Firefox)
* Native English speaker
* 18 to 35 years old

Exclusion Criteria:

* Planning to be without Internet access during the scheduled intervention time

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale | Baseline and 3 weeks

SECONDARY OUTCOMES:
Emotion Regulation Questionnaire | Baseline and 3 weeks
Perseverative Thinking Questionnaire | Baseline and 3 weeks
Subjective Happiness Scale | Baseline and 3 weeks
Positive and Negative Affect Schedule | Baseline and 3 weeks
Utilization and Attrition | Baseline-week 3
  activity level (word count, number of social actions, average number and length of web sessions)

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind W Picard, Sc.D, Principal Investigator — Massachusetts Institute of Technology

REFERENCES:
- [Derived] Morris RR, Schueller SM, Picard RW. Efficacy of a Web-based, crowdsourced peer-to-peer cognitive reappraisal platform for depression: randomized controlled trial. J Med Internet Res. 2015 Mar 30;17(3):e72. doi: 10.2196/jmir.4167. PMID 25835472